CLINICAL TRIAL: NCT04575259
Title: Open Label Extension Study for Patients With Parkinson's Disease With Dementia Enrolled in Study ANAVEX2-73-PDD-001
Brief Title: OLE Study for Patients With Parkinson's Disease With Dementia Enrolled in Study ANAVEX2-73-PDD-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: Anavex Australia Pty Ltd. (Industry); Anavex Germany GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANAVEX2-73-PDD-EP-001
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease Dementia
MeSH Terms: interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ANAVEX2-73 Active (Experimental): Oral capsules
  Interventions: Drug: ANAVEX2-73

INTERVENTIONS:
Drug: ANAVEX2-73 — Oral capsules
  Other Names: Blarcamesine

SUMMARY:
This is a Phase 2 open-label extension study to evaluate the effects of ANAVEX2-73 on safety and efficacy of daily treatment.

DETAILED DESCRIPTION:
This is a Phase 2 open-label extension study to evaluate the effects of ANAVEX2-73 on safety and efficacy of daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous completion of participation in the ANAVEX2-73-PDD-001 study.
* Caregivers and subjects (or legal representative) must understand and have signed approved informed consent.
* Caregivers and subjects (or legal representative) must be able to understand study requirements and be willing to follow instructions.
* Stable regimen of anti-Parkinson's disease medications (including levodopa, dopamine agonists, MAO-B inhibitors, or the COMT inhibitor entacapone), which has been stable for at least 4 weeks prior to Baseline.
* Treatment with cholinesterase inhibitor (rivastigmine, donepezil and galantamine (Exelon®, Aricept®, or Reminyl®) will be permitted, provided the dose has been stable for a minimum of 8 weeks prior to joining this study.
* Subjects with history of depression on antidepressant medications will be allowed if depression is controlled and they have been on a stable daily dose of the antidepressant for ≥8 weeks before Baseline.
* Contraception: Women of childbearing potential must use an acceptable method of contraception starting 4 weeks prior to study drug administration and for a minimum of 4 weeks after study completion. Otherwise, women must be postmenopausal (at least one year absence of vaginal bleeding or spotting) as confirmed by FSH greater than or equal to 40 mIU/mL or 40 IU/L or be surgically sterile.
* Men with a potentially fertile partner must have had a vasectomy or be willing to use an acceptable method of contraception for the duration of the study and for 3 months after study drug discontinuation.

Exclusion Criteria:

* History of any significant neurologic or psychiatric disorder other than PD that can contribute to cognitive impairment.
* Any other condition or clinically significant abnormal findings on the physical or neurological examination, medical and psychiatric history, at screening or at baseline that, in the opinion of the Investigator, would make the subject unsuitable for the study.
* Potential symptomatic causes of cognitive impairment including but not limited to
* abnormal thyroid function test at screening (TSH)
* abnormal B12 level at screening
* MRI findings (by history) pointing to a potential symptomatic cause of cognitive dysfunction, including significant vascular changes, or communicating hydrocephalus.
* Treatment with memantine or amantadine. If appropriate the drugs can be discontinued for a minimum of 4 weeks prior to enrollment.
* History of depression as measured by Beck Depression Inventory score >17 at screening.
* Treatment with any other investigational drug or device within 4 weeks prior to screening.
* Smoking > 1 pack of cigarettes per day (as assessed for the 4 weeks prior to screening).
* Women who are pregnant or lactating.
* Known allergy or sensitivity to ANAVEX2-73 or any of its components.
* Suicidal ideation on the Columbia Suicide Severity Rating Scale (C-SSRS) of type 4 or type 5, or any suicidal behavior, in the past 6 months. Type 4 indicates active suicidal ideation with some intent to act, without a specific plan. Type 5 indicates active suicidal ideation with a specific plan and intent.
* Use of centrally acting anticholinergic drugs during the 4 weeks before enrollment.
* Medications used for overactive bladder will be allowed provided that the regimen has been stable 4 weeks prior to enrollment.
* Treatment with any dopamine receptor blocking medications with the exception of low dose quetiapine (≤50 mg/day). Pimavanserin (≤34 mg/day) will be allowed.
* History of neurosurgical intervention (e.g., deep brain stimulation) for PD.
* Unpredictable motor fluctuations that would interfere with administering cognitive assessments in the ON state.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 48 weeks
  To continue assessing the safety and tolerability of ANAVEX2-73

SECONDARY OUTCOMES:
RSBDQ (REM Sleep Behavior Disorder Screening Questionnaire) | 48 weeks
  Change from baseline to End of Treatment as measured by RSBDQ
MDS-UPDRS Part III Total Score (Motor Scores) | 48 weeks
  Change from baseline to End of Treatment as measured by MDS-UPDRS Part III Total Score (Motor Scores)
MoCA (Montreal Cognitive Assessment) | 48 weeks
  Change from baseline to End of Treatment as measured by MoCA

OTHER OUTCOMES:
Microbiota | 48 weeks
  Change from baseline to End of Treatment as measured by microbiota

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (2):
  - KaRa MINDS, Macquarie Park, New South Wales
  - Hammond Care, Malvern, Victoria
- Spain (8):
  - Hospital Mutua Terrasa, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital del Henares, Coslada
  - Clínica Universidad de Navarra (CUN) - Sede Madrid- Servicio de Neurología -, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitario Virgen del Rocío, Seville